CLINICAL TRIAL: NCT04749927
Title: Prediction of Incident Atherosclerotic Cardiovascular Disease From Retinal Photographs Via Deep Learning
Brief Title: Deep Learning of Retinal Photographs and Atherosclerotic Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0951
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research team has developed a deep learning algorithm that predicts anthropometric factors from fundus photographs and an algorithm that predicts cardiovascular disease risk. Fundus photographs are taken for various cardiovascular diseases (myocardial infarction, heart failure, hypertension with target organ damage, high-risk dyslipidemia, diabetic patients, and low-risk hypertension patients), and a deep learning algorithm for predicting developed anthropometric factors will be validated. Fundus photographs will also be taken twice in the first year, and additional fundus photographs will be taken two years later. Major cardiovascular events will be followed up for 5 years to verify the deep learning algorithm predicting cardiovascular disease risk prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Myocardial infarction (Patients diagnosed with myocardial infarction within 5 years and confirmed significant coronary artery stenosis by cardiovascular angiography)
2. Heart failure with reduced EF (<40% of LVEF on echocardiography or magnetic resonance imaging)
3. Heart failure with preserved EF (≥40% of LVEF on echocardiography and NT-proBNP ≥200 pg/mL and LAVI ≥ 34 ml/m2 or LVMI ≥115 g/m2 (men) or LVMI ≥95 g/m2 (women))
4. High risk subclinical atherosclerosis (no symptom and ≥50% stenosis of coronary artery on coronary angio CT or asymptomatic PAOD or cerebral aneurysm or ≥50% stenosis of cerebral artery or ABI <0.9 or ≥2mm of atherosclerotic plaque or hypoechogenic plaque on carotid ultrasound)
5. Hypertension with target organ damage (proteinuria [urine albumin/creatinine ratio ≥ 30 mg/g or protein/creatinine ratio ≥ 150 mg/g or 24 hour urine albumin ≥30mg/day or 24 hour urine protein ≥ 150mg/day] or LV hypertrophy [on EKG or echocardiography] or cfPWV > 10 m/sec or baPWV > 1800 cm/sec or eGFR < 60 ml/min/1.72 m2 or atherosclerotic cardiovascular disease or white matter hyperintensity on brain MRI)
6. High risk dyslipidemia (LDL-cholesterol >190 mg/dL or > 160 mg/dL inspire of use of moderate or high intensity statin)
7. Diabetes (Type 2 diabetes with more than 5 years of diagnosis or type 1 diabetes with more than 10 years of diagnosis)
8. Low risk (Hypertension that does not meet the above criteria and is controlled by 3 drugs or less 2) Dyslipidemia that does not meet the above criteria and is controlled below the target LDL)

Exclusion Criteria:

1. Serious eye diseases that make it impossible to take adequate quality fundus photography
2. If the subject cannot read and sign the consent form in person

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visiting outpatient clinic in the tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2029-10-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular disease | 4 years
  Composite of myocardial infarction, stroke, coronary revascularization including percutaneous coronary intervention and coronary bypass graft, and hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Sungha Park, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No